CLINICAL TRIAL: NCT00119392
Title: A Phase II Trial Evaluating the Safety and Efficacy of Non-myeloablative 90Y-Ibritumomab Tiuxetan (Anti-CD20) Antibody With Fludarabine, Low-Dose Total Body Irradiation (TBI) and HLA Matched Allogeneic Transplantation for Relapsed B-cell Lymphoma
Brief Title: Yttrium Y 90 Ibritumomab Tiuxetan, Fludarabine, Radiation Therapy, and Donor Stem Cell Transplant in Treating Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ajay Gopal, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1726.00; NCI-2010-01381 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2005-07-12; First posted 2005-07-13 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Splenic Marginal Zone Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia | interventions — Rituximab; Cyclosporine; fludarabine phosphate; Mycophenolic Acid; ibritumomab tiuxetan; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (90Y ibritumomab tiuxetan, hematopoietic transplant) (Experimental): See Detailed Description
  Interventions: Biological: rituximab; Drug: cyclosporine; Drug: fludarabine phosphate; Drug: mycophenolate mofetil; Radiation: yttrium Y 90 ibritumomab tiuxetan; Procedure: peripheral blood stem cell transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Radiation: total-body irradiation

INTERVENTIONS:
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: cyclosporine — Given orally
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: mycophenolate mofetil — Given orally
  Other Names: Cellcept; MMF
Radiation: yttrium Y 90 ibritumomab tiuxetan — Given IV
  Other Names: 90Y ibritumomab tiuxetan; IDEC Y2B8; Y90 Zevalin; Y90-labeled ibritumomab tiuxetan
Procedure: peripheral blood stem cell transplantation — Undergo transplantation
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo transplantation
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI

SUMMARY:
Monoclonal antibodies, such as yttrium Y 90 ibritumomab tiuxetan, can block find cancer cells and either kill them or carry cancer-killing substances to them without harming normal cells. Giving monoclonal antibodies, low doses of chemotherapy, such as fludarabine phosphate, and low dose total-body radiation therapy before a donor peripheral stem cell transplant helps stop the growth of cancer cells and also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine or mycophenolate mofetil after the transplant may stop this from happening

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility, safety, and potential efficacy of treating patients with B-Cell non-Hodgkin lymphoma (NHL) with 90Y-ibritumomab tiuxetan, combined with HLA-matched related or unrelated donor hematopoietic cell transplantation.

OUTLINE: Patients receive rituximab intravenously (IV) followed by, no more than 4 hours later, indium In 111 ibritumomab tiuxetan (for imaging) IV over 10 minutes on day -21. Patients undergo gamma camera imaging on day -19. Patients receive rituximab IV followed by, no more than 4 hours later, yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes on day -14. Patients also receive fludarabine phosphate IV over 30-60 minutes on days -7 to -5 and undergo low-dose total-body irradiation (TBI) on day 0. After TBI, patients undergo allogeneic peripheral blood stem cell transplantation (PBSCT) on day 0. Patients who undergo PBSCT from a related donor receive oral cyclosporine twice daily on days -3 to 56 followed by a taper to day 180 in the absence of graft-versus-host disease (GVHD). These patients also receive oral mycophenolate mofetil twice daily on days 0 to 27. Patients who undergo PBSCT from an unrelated donor receive oral cyclosporine twice daily on days -3 to 100 followed by a taper over 11 weeks in the absence of GVHD. These patients also receive oral mycophenolate mofetil three times daily on days 0 to 40 followed by a taper to day 96.

After completion of study treatment, patients are followed up at 1, 3, 6, and 12 months, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of a lymphoid malignancy expressing the cluster of differentiation (CD)20 antigen and have failed at least one prior standard systemic therapy
* Patients must have evidence of persistent lymphoma by physical examination, radiographic studies, bone marrow evaluation, flow cytometry, or polymerase chain reaction (PCR)
* Creatinine < 2.0
* Bilirubin < 1.5 mg/dL
* Patients must have an expected survival of > 60 days and must be free of major infection including human immunodeficiency virus (HIV)
* Patients must have an HLA-identical related or unrelated donor
* DONOR: Donor eligibility includes both HLA-matched relatives or HLA matched, unrelated volunteer donors; related donors should be matched by molecular methods at the intermediate resolution level at HLA-A, B, C, and DRB1 according to FHCRC Standard Practice Guidelines and to the allele level at DQB1; unrelated donors should be identified using matching criteria that follows the FHCRC Standard Practice Guidelines limiting the study to eligible donors that are allele matched for HLA-A, B, C, DRB1, and DQB1 (Grade1), and accepting up to one allele mismatch as per Standard Practice Grade 2.1 for HLA-A, B, or C
* Donor must consent to granulocyte colony-stimulating factor (G-CSF) (filgrastim) administration and leukapheresis
* Donor must have adequate veins for leukapheresis or agree to placement of central venous catheter (femoral, subclavian)

Exclusion Criteria:

* Systemic anti-lymphoma therapy given in the previous 30 days
* Patients who have experienced progressive disease within 3 months of prior Bexxar or Zevalin
* Inability to understand or give an informed consent
* Central nervous system lymphoma
* Pregnancy
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Southwest Oncology Group (SWOG)/Eastern Cooperative Oncology Group (ECOG) performance score > 2
* Eligible for radioimmunotherapy-based autologous transplant trial
* Medical condition that would contraindicate allogeneic transplantation
* Evidence of Human Anti-Mouse Antibody (HAMA) for patients with prior exposure to therapeutic murine antibodies
* Eligible for other therapeutic options that will be more likely to have a better long-term disease-free survival with lower potential toxicity (e.g., non-transplant therapy, autologous transplants, etc.) than this study
* Other grave medical conditions considered to represent contraindications to bone marrow transplant (BMT) (e.g. unstable angina, pulmonary dysfunction [diffusing capacity of the lung for carbon monoxide (DLCO) < 30%, total lung capacity (TLC) < 30%, continuous supplemental oxygen], acquired immune deficiency syndrome [AIDS], etc.)
* DONOR: Identical twin
* DONOR: Age less than 12 years
* DONOR: Pregnancy
* DONOR: Infection with HIV
* DONOR: Inability to achieve adequate venous access
* DONOR: Known allergy to G-CSF
* DONOR: Current serious systemic illness or infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-06; Primary Completion 2009-07 (Actual); Study Completion 2016-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Gopal, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Puronen CE, Cassaday RD, Stevenson PA, Sandmaier BM, Flowers ME, Green DJ, Maloney DG, Storb RF, Press OW, Gopal AK. Long-Term Follow-Up of 90Y-Ibritumomab Tiuxetan, Fludarabine, and Total Body Irradiation-Based Nonmyeloablative Allogeneic Transplant Conditioning for Persistent High-Risk B Cell Lymphoma. Biol Blood Marrow Transplant. 2018 Nov;24(11):2211-2215. doi: 10.1016/j.bbmt.2018.06.033. Epub 2018 Jul 3. PMID 30454872
- [Derived] Gopal AK, Guthrie KA, Rajendran J, Pagel JM, Oliveira G, Maloney DG, Matesan MC, Storb RF, Press OW. (9)(0)Y-Ibritumomab tiuxetan, fludarabine, and TBI-based nonmyeloablative allogeneic transplantation conditioning for patients with persistent high-risk B-cell lymphoma. Blood. 2011 Jul 28;118(4):1132-9. doi: 10.1182/blood-2010-12-324392. Epub 2011 Apr 20. PMID 21508413

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (90Y Ibritumomab Tiuxetan, Hematopoietic Transplant)
Started | 45
Completed | 40
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (90Y Ibritumomab Tiuxetan, Hematopoietic Transplant)
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 58 [29 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Treatment Related Mortality (TRM)
Description: Cumulative incidence rate of treatment related mortality with relapse as a competing risk, assessed at 30 months.
Time Frame: At day +100
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Treatment (90Y Ibritumomab Tiuxetan, Hematopoietic Transplant)
Number analyzed (Participants) | 40
percent | 16 [4 to 28]

2. Secondary Outcome: Overall and Progression-free Survival
Description: Kaplan-Meier estimates for overall survival (OS) and progression free survival (PFS) assessed at two years.
Time Frame: Up to 8 years
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Treatment (90Y Ibritumomab Tiuxetan, Hematopoietic Transplant)
Number analyzed (Participants) | 40
percent
  Overall survival | 54 [37 to 68]
  Progression free survival | 31 [16 to 48]

3. Secondary Outcome: Response Rates
Time Frame: Up to 8 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (90Y Ibritumomab Tiuxetan, Hematopoietic Transplant)
Number analyzed (Participants) | 42
Participants | 25

4. Secondary Outcome: Engraftment and Hematopoietic Toxicity
Description: Median number of days after transplantation to a neutrophil count less than 500 neutrophils per microliter and a platelet count less than 50,000 platelets per microliter.
Time Frame: At day +100
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (90Y Ibritumomab Tiuxetan, Hematopoietic Transplant)
Number analyzed (Participants) | 40
days
  Neutrophils | 17 [0 to 34]
  Platelets | 11 [0 to 147]

5. Secondary Outcome: Incidence and Severity of Acute Graft-versus-host Disease (GVHD) and Chronic GVHD.
Time Frame: At day +84
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (90Y Ibritumomab Tiuxetan, Hematopoietic Transplant)
Number analyzed (Participants) | 40
Participants
  Acute GVHD: Grade 1-2 | 27
  Acute GVHD: Grade 3 | 4
  Chronic extensive GVHD | 5

ADVERSE EVENTS:
Arm/Group | Treatment (90Y Ibritumomab Tiuxetan, Hematopoietic Transplant)
Serious Adverse Events (participants affected / at risk) | 8/40
Other Adverse Events (participants affected / at risk) | 36/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (90Y Ibritumomab Tiuxetan, Hematopoietic Transplant) (N=40)
Neutropenic fever (Blood and lymphatic system disorders) | 1
Bone pain (General disorders) | 2
Renal insufficiency (Renal and urinary disorders) | 1
Hypotension (Vascular disorders) | 1
Stroke (Nervous system disorders) | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1
Sepsis (Infections and infestations) | 1
Disease progression (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (90Y Ibritumomab Tiuxetan, Hematopoietic Transplant) (N=40)
Anorexia (Metabolism and nutrition disorders) | 9
Arrhythmia (Cardiac disorders) | 3
Infection (Infections and infestations) | 27
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 5
Diarrhea (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 8
Neutropenia (Blood and lymphatic system disorders) | 26
Thrombocytopenia (Blood and lymphatic system disorders) | 23
Febrile Neutropenia (Blood and lymphatic system disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 11
Pain (General disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hypertension (Vascular disorders) | 9
Hypotension (Vascular disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 7
Leukopenia (Blood and lymphatic system disorders) | 12
Lymphopenia (Blood and lymphatic system disorders) | 21
Nausea (Gastrointestinal disorders) | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Elevated ALT (Investigations) | 2
Elevated Creatinine (Investigations) | 2
Decreased WBC (Investigations) | 5
Hyponatremia (Metabolism and nutrition disorders) | 4
Neuropathy (Nervous system disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Hypophosphatemia (Gastrointestinal disorders) | 2
Edema (General disorders) | 3
Insomnia (Psychiatric disorders) | 2
Decreased hemoglobin (Investigations) | 2
Embolism Thrombosis/Thrombus (Vascular disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Obstruction (Gastrointestinal disorders) | 3
Weakness (General disorders) | 2
Osteopenia (Musculoskeletal and connective tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes